CLINICAL TRIAL: NCT03190044
Title: A Fixed Combination of Magnesium, Partenium, Andrographis, Co-enzyme Q10 and Riboflavin (PACR) as Prophylactic Treatment for Migraine: a Randomized Controlled Double Blind Study (ParMig Study)
Brief Title: Magnesium, Partenium, Andrographis, Co-enzyme Q10 and Riboflavin (PACR) in Migraine Prophylaxis
Acronym: ParMig
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Gianluca Coppola (Unknown); Francesco Pierelli (Unknown)
Responsible Party: Principal Investigator, Cherubino DI LORENZO, Research Fellow, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ParMig Study
Record Dates: First submitted 2017-06-06; First posted 2017-06-16 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Placebo and 'verum' pills have the similar shape and colour.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Migraineurs (verum) (Experimental): One pill per day of PACR: magnesium 281,25 mg; partenium 150 mg (partenolides 1200mcg); andrographis 100 mg (andrographolides 10 mg); co-enzyme Q10 20 mg; riboflavin 4,8 mg.
  Interventions: Dietary Supplement: PACR
- Migranineurs (placebo) (Placebo Comparator): One pill per day of placebo: Cellulose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: PACR — Daily assumption of PACR for a 3-month period
  Arms: Migraineurs (verum)
Dietary Supplement: Placebo — Daily assumption of placebo
  Arms: Migranineurs (placebo)

SUMMARY:
Migraine is a highly disabling disorder that affects hundreds of millions of people around the world. Yet, a little number of prophylactic treatments are available still now. The limited number of available drugs leads to a wide use of nutraceutical compounds in migraine therapy. To improve the efficacy, some of these nutraceuticals were combined. So far, we do not know if these combinations are really more effective than the single compounds alone, or an anti-synergic effect could be present because of a reciprocal antagonism of effects. For this reason, we decided to test the efficacy of a fixed combination of magnesium, partenium, andrographis, co-enzyme Q10 and riboflavin (PACR) as prophylactic treatment for migraine in a randomized controlled double blind study.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of migraine (with or without aura)
* both genders
* age between 18 and 65 y.o.
* more than 1 year of migraine history
* no other headache conditions
* a migraine frequency between 2 and 8 per month

Exclusion Criteria:

* Prophylactic treatments in the last 3 months
* pregnancy or lactation
* other medical conditions that requires a daily drug assumption
* intolerance or allergic reactions to some of compounds of the product.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2017-06-06 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Migraine improvement in terms of responder rate | 3 months
  Number of subjects that at least have a reduction of 50% in terms of migraine frequency

SECONDARY OUTCOMES:
Migraine improvement in terms of frequencies | 3 months
  reduction of migraine in terms of number of attacks, headache days, and number of analgesics per month.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Pierelli, MD, Study Chair — University of Roma La Sapienza
Locations (1):
- Policlinico Umberto I, Rome, Italy

IPD SHARING:
Plan to Share IPD: No